CLINICAL TRIAL: NCT06339970
Title: Effects of Slider Versus Tensioners Nerve Gliding Technique Along With Mulligan Spinal Mobilization on Pain, Range of Motion and Disability in Patients With Cervical Radiculopathy.
Brief Title: Effects of Slider Versus Tensioners Nerve Gliding in Cervical Radiculopathy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0199 iram
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Cervical Radiculopathy
Keywords: Tensioners mobilization, Manual Therapy and neck pain
MeSH Terms: conditions — Radiculopathy; Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slider Nerve Gliding Technique along with Mulligan Spinal Mobilization Technique (Active Comparator): Therapist approaches the desired level of spinous process from medial aspect of the thumb of one hand which is reinforced by the index finger of the other hand. Second therapist places his axilla over the patient's shoulder to add shoulder depression component. The second therapist performs components of the nerve to be test one by one (distal to proximal or proximal to distal sequence) depending upon patient's offending movements and painful range.Pure transverse glide is performed from affected to unaffected side. While the glide is sustained, another therapist mobilizes the median nerve by performing desired neurodynamic sliding movement. Apply this protocol for 4 weeks 12 Sessions (3 sessions in a week) and 10 sec rest between each segment, 3 sets of 10 repetitions.
  Interventions: Other: Slider Nerve Gliding Technique along with Mulligan Spinal Mobilization Technique
- Tensioners Nerve Gliding Technique along with Mulligan Spinal Mobilization Technique (Experimental): Therapist approaches the desired level of spinous process from medial aspect of the thumb of one hand which is reinforced by the index finger of the other hand. Second therapist places his axilla over the patient's shoulder to add shoulder depression component. The second therapist performs components of the nerve to be test one by one (distal to proximal or proximal to distal sequence) depending upon patient's offending movements and painful range.Pure transverse glide is performed from affected to unaffected side. While the glide is sustained, another therapist mobilizes nerve by performing desired neurodynamic gliders movement and progressing to tensioners. Apply this protocol for 4 weeks 12 Sessions (3 sessions in a week) and 10 sec rest between each segment, 3 sets of 10 repetitions.
  Interventions: Other: Tensioners Nerve Gliding Technique along with Mulligan Spinal Mobilization Technique

INTERVENTIONS:
Other: Slider Nerve Gliding Technique along with Mulligan Spinal Mobilization Technique — In this group 21 patients will perform Slider Nerve Gliding Technique along with Mulligan Spinal Mobilization Technique.Protocol for 4 weeks 12 Sessions (3 sessions in a week) and 10 sec rest between each segment, 3 sets of 10 repetitions. Patient is sitting in the chair / plinth. Therapist's standing behind the patient.
  Arms: Slider Nerve Gliding Technique along with Mulligan Spinal Mobilization Technique
Other: Tensioners Nerve Gliding Technique along with Mulligan Spinal Mobilization Technique — In this group 21 patients will perform Tensioners Nerve Gliding Technique along with Mulligan Spinal Mobilization Technique.Protocol for 4 weeks 12 Sessions (3 sessions in a week) and 10 sec rest between each segment, 3 sets of 10 repetitions. Patient is sitting in the chair / plinth. Therapist's standing behind the patient.
  Arms: Tensioners Nerve Gliding Technique along with Mulligan Spinal Mobilization Technique

SUMMARY:
This study will be a randomized clinical trial in which Slider versus Tensioners Nerve Gliding Technique along with Mulligan Spinal Mobilization will be applied on the individuals with cerviculorediculopathy and changes will be recorded using different methods and tools. Convenient sampling technique will be used to collect the data. The sample size of 40 patients will be recruited. Patients will be randomly allocated into two different groups through sealed envelope method.20 patients will be allocated in each group A will be treated with Slider Nerve Gliding Technique along with Mulligan Spinal Mobilization Technique; Group B will be treated with Tensioners Nerve Gliding Technique along with Mulligan Spinal Mobilization Technique .Numeric Pain Rating Scale (NPRS), Neck Disability Index (NDI) and goniometer will be used as Data collecting tools. After data collection from defined study setting, data will be entered and analyzed.

DETAILED DESCRIPTION:
Neck pain is widespread and causes significant pain and disability. In the setting of cervical radiculopathy, because the nerve root of a spinal nerve is compressed It is frequently caused by cervical disc herniation and cervical spondylitis. Compression can result from intervertebral disc herniation, osteophyte formation, or other mass effects near the exit foramen of the cervical spine. This results in lower motor neurons symptoms and often presents with arm pain, weakness, and/or sensory loss, with or without associated neck pain. The most common causes of cervical radiculopathy are cervical disc herniation and cervical spondylosis.

The main aim of our study to determine which combination of techniques Slider versus Tensioners Nerve Gliding Technique along with Mulligan Spinal Mobilization is more effective on Pain, Range of Motion and Disability in patients with Cervical Radiculopathy.

Combination of mulligan mobilization with slider and tensioners techniques to determine which combination of technique is more helpful in reducing overall disease burden and will help in increasing Quality of life.Bothcombination combination are checked individually before but their effects are not compared previously.

ELIGIBILITY:
Inclusion Criteria: • Patient with cervical radiculopathy

* Both gender Age
* Participants having range 20-60 years both male and female are included.
* Unilateral neck pain refers to upper extremity from 2-3 weeks.
* Positive upper limb tension test, spurling test, cervical distraction test and ipsilateral cervical rotation less than 60.
* NDI less than 50%
* NPRS less than 3 more than 7

Exclusion Criteria:

* Inflammation malignancy, neurological disorder
* Metabolic disorders
* Neck pain associated with headache and facial pain
* VBI, vertigo, dizziness, motor imbalance, vertebral impairment, pregnancy, skin allergy
* History of recent surgery, trauma and fractures of cervical spine, dislocation, subluxation of upper limb,
* rheumatoid arthritis, osteoporosis, spondylolistheasis, cervical surgeries skin allergy, referred pain in patient with cardiac ischemia
* Patients having any other therapeutic intervention or medical treatment

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4 Weeks
  NPRS consists of a scale with 0-10 readings. The zero denotes no pain while 1, 2, 3 denotes to mild pain, 4, 5, 6 denotes to moderate pain while 7-10 denotes to severe pain.
Neck disability index | 4 Weeks
  .The NDI consists of ten questions. Each question has six different assertions expressing progressive levels of pain or limitation in activities. Item scores range from 0 (no pain or limitation) to 5 (as much pain as possible or maximal limitation). The total NDI score ranges from 0 to 5 points. Higher scores indicate greater disability.
Goniometer | 4 Weeks
  Active Range of Motion of the patient will be assessed using a universal standard goniometer for cervical flexion, extension, side flexion (left and right), rotation (left and right). The data will be collected at baseline cervical goniometry.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad sanaullah, MS, Principal Investigator — Riphah International University
Locations (1):
- Sehat Medical Compolex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCartney S, Baskerville R, Blagg S, McCartney D. Cervical radiculopathy and cervical myelopathy: diagnosis and management in primary care. Br J Gen Pract. 2018 Jan;68(666):44-46. doi: 10.3399/bjgp17X694361. No abstract available. PMID 29284641
- [Background] Margetis K, Magnus W, Mesfin FB. Cervical Radiculopathy. 2025 Aug 6. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK441828/ PMID 28722858
- [Background] Carroll LJ, Hogg-Johnson S, van der Velde G, Haldeman S, Holm LW, Carragee EJ, Hurwitz EL, Cote P, Nordin M, Peloso PM, Guzman J, Cassidy JD; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Course and prognostic factors for neck pain in the general population: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S75-82. doi: 10.1097/BRS.0b013e31816445be. PMID 18204403
- [Background] Sharma S, Balthillaya G, Rao R, Mani R. Short term effectiveness of neural sliders and neural tensioners as an adjunct to static stretching of hamstrings on knee extension angle in healthy individuals: A randomized controlled trial. Phys Ther Sport. 2016 Jan;17:30-7. doi: 10.1016/j.ptsp.2015.03.003. Epub 2015 Mar 17. PMID 26482098
- [Background] Papacharalambous C, Savva C, Karagiannis C, Giannakou K. The effectiveness of slider and tensioner neural mobilization techniques in the management of upper quadrant pain: A systematic review of randomized controlled trials. J Bodyw Mov Ther. 2022 Jul;31:102-112. doi: 10.1016/j.jbmt.2022.03.002. Epub 2022 Mar 18. PMID 35710209
- [Background] Coppieters MW, Butler DS. Do 'sliders' slide and 'tensioners' tension? An analysis of neurodynamic techniques and considerations regarding their application. Man Ther. 2008 Jun;13(3):213-21. doi: 10.1016/j.math.2006.12.008. Epub 2007 Mar 30. PMID 17398140
- [Background] Shafique S, Ahmad S, Shakil-Ur-Rehman S. Effect of Mulligan spinal mobilization with arm movement along with neurodynamics and manual traction in cervical radiculopathy patients: A randomized controlled trial. J Pak Med Assoc. 2019 Nov;69(11):1601-1604. doi: 10.5455/JPMA.297956.. PMID 31740863
- [Background] Michener LA, Snyder AR, Leggin BG. Responsiveness of the numeric pain rating scale in patients with shoulder pain and the effect of surgical status. J Sport Rehabil. 2011 Feb;20(1):115-28. doi: 10.1123/jsr.20.1.115. PMID 21411827
- [Background] Young IA PT, DSc, Dunning J PT, DPT, Butts R PT, PhD, Mourad F PT, DPT, Cleland JA PT, PhD. Reliability, construct validity, and responsiveness of the neck disability index and numeric pain rating scale in patients with mechanical neck pain without upper extremity symptoms. Physiother Theory Pract. 2019 Dec;35(12):1328-1335. doi: 10.1080/09593985.2018.1471763. Epub 2018 Jun 1. PMID 29856244
- [Background] Jorritsma W, Dijkstra PU, de Vries GE, Geertzen JH, Reneman MF. Detecting relevant changes and responsiveness of Neck Pain and Disability Scale and Neck Disability Index. Eur Spine J. 2012 Dec;21(12):2550-7. doi: 10.1007/s00586-012-2407-8. Epub 2012 Jul 3. PMID 22752592
- [Background] Farooq MN, Mohseni Bandpei MA, Ali M, Khan GA. Reliability of the universal goniometer for assessing active cervical range of motion in asymptomatic healthy persons. Pak J Med Sci. 2016 Mar-Apr;32(2):457-61. doi: 10.12669/pjms.322.8747. PMID 27182261